CLINICAL TRIAL: NCT03466138
Title: Performance Assessment of the Physiological Monitoring Device - PMD-200 - in Subjects Requiring Surgery Under General Anesthesia
Brief Title: Performance Assessment of the PMD-200 in Subjects Requiring Surgery Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Medasense Biometrics Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: CLI-16-02
Record Dates: First submitted 2017-12-27; First posted 2018-03-15 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General Anesthesia: subjects requiring a surgical procedure under general anesthesia. monitored by PMD-200
  Interventions: Device: PMD-200

INTERVENTIONS:
Device: PMD-200 — The PMD-200 system is comprised of a console and designated finger probe with 4 sensors. The Sensors are Photoplethysmography (PPG) Galvanic Skin Response (GSR), Accelerometer (ACC) and Thermistor (TMP)

SUMMARY:
The proposed study is designed to further demonstrate the performance of the Nociception Level (NoL) Index - in surgical patient under general anesthesia, by evaluating its response to controlled changes in the levels of noxious stimuli/analgesia and to correlate early outcome predictors to the NoL values throughout the surgical procedure, thus provide the medical caregiver general recommendations on how to interpret the NoL Index in terms of magnitude and direction, and how to utilize it during the surgical procedure.

DETAILED DESCRIPTION:
The proposed study is designed to further demonstrate the performance of the NoL Index in surgical patient under general anesthesia, by evaluating its response to controlled changes in the levels of noxious stimuli/analgesia mentioned characteristics and to correlate early outcome predictors to the NoL values throughout the surgical procedure, thus provide the medical caregiver general recommendations on how to interpret the NoL Index in terms of magnitude and direction, and how to utilize it during the surgical procedure.

In this study the investigators plan to demonstrate that the NoL Index is a continuous index. It is anticipated that a higher level of nociception will correspond to a higher NoL index. On the other hand, it is anticipated that higher levels of analgesic agent for the same noxious stimulus will lead to a lower NoL index. This will be achieved by measuring the NoL response to various types of noxious stimuli, varying in their intensities, under different levels of analgesic agents.

The noxious stimuli that will be used in this pivotal study are:

1. - Intubation
2. - Incision and/or trocar insertion
3. - Internal handling during the surgical procedure
4. - Extubation
5. - Other specific pain event related to the surgical procedure (e.g. bone related treatment in orthopedic, muscle tension or cut etc.).

The study population includes subjects requiring a surgical procedure under general anesthesia. During the surgical procedure the subject is anesthetized (by various anesthetic agents) and paralyzed (by muscle relaxant agents). Thus, the response to noxious stimuli under those conditions will be related to the underlying physiological response. The participants will be monitored, as in a typical surgery and according to the local guidelines, by various types of monitoring devices, such as: vital signs, pulse oximeter, Bispectral Index (BIS), Electroencephalography (EEG) etc. Therefore, patients suffering from fluctuations in their vital signs and hemodynamic parameters during the surgical procedure, can be detected by the various monitors. However, assessment of the level of nociception is still complex, subjective and mainly depends on the physician's experience and knowledge.

Development of a nociception monitor that may present an index to assess the level of nociception will allow the anesthesiologist better patient management during the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* The subject age is > 18 years old
* The subject requires surgery under general anesthesia.
* A blood pressure measurement (via arterial line or cuff) will be available during the surgical procedure.
* The subject signed an Informed Consent Form (ICF)

Exclusion Criteria:

* History of severe cardiac arrhythmias within the last 12 months
* Pregnancy or lactation
* Chronic pain conditions or analgesic usage (> 1 month of large doses of opioids: more than 30mg PO equivalent of morphine)

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects requiring a surgical procedure under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
demonstrate the NoL Index correlation prior and following a noxious stimuli. | Through study completion, about one year
  The primary objective is to demonstrate the NoL Index is correlates with changes in the nociception levels of the subject during the surgical procedure prior and following a noxious stimuli.

SECONDARY OUTCOMES:
Correlation between the NoL Index and other nociception predictors (such as heart rate - Beats per Minute) following a noxious stimuli. | Through study completion, about one year
  The NoL values can be correlate to other nociception predictors (e.g heart rate, blood pressure) following a noxious stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Tibi Ezri, Prof., Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Holon, Israel